CLINICAL TRIAL: NCT05556564
Title: The Impact of Migraine on Canadians' Productivity: A Real-World Pharmacy-Based Study
Status: Completed | Type: Observational
Sponsor: PeriPharm (Other)
Responsible Party: Sponsor
Other Study IDs: PROxy202201
Record Dates: First submitted 2022-09-20; First posted 2022-09-27 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Observation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No group
  Interventions: Drug: observational study

INTERVENTIONS:
Drug: observational study — No intervention, observational study

SUMMARY:
This is a cross-sectional, real-world observational, community pharmacy-based study in which adults treated with a triptan for their migraine will self-report productivity and activity impairment using a web-based portal or paper-based questionnaire.

DETAILED DESCRIPTION:
The primary objective of this study is to estimate the productivity and activity impairment associated with migraine in adults treated with a triptan.

Participant identification will be made using pharmacies member of the PROxy Network. Eligible participants will be identified using the prescription of any formulation of triptans either when filling or refilling a prescription of a triptan or in the pharmacy electronic database (patients with a renewal in the last 3 months).

The PROxy Network is a research network bringing together community pharmacies across Quebec to facilitate the generation of real-world evidence. This network is designed to better understand a disease or a treatment using patient-reported outcomes (PROs). The PROxy Network is an initiative of PeriPharm Inc., a company specializing in pharmacoeconomics and outcomes research.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* New or current prescription (renewal in the last 3 months) of any formulation of triptans medication (i.e., almotriptan, eletriptan, naratriptan, rizatriptan, sumatriptan, zolmitriptan and frovatriptan);
* Working full or part-time or going to school full or part-time;
* Ability to read and understand English or French;
* Signature of informed consent form (ICF).

Exclusion Criteria:

* Patients participating in a clinical trial.
* Patients filling a one-time vacation/emergency prescription (i.e. without a complete pharmacy file).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with migraine treated with triptans in Canada
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
The Migraine Disability Assessment (MIDAS) questionnaire | Baseline
  Patient-reported outcome: The Migraine Disability Assessment (MIDAS) is a 5-item, self-administered questionnaire designed to quantify headache-related disability over the past 3 months. The MIDAS is scored as the sum of five questions, each measured as days in the last 3 months, and then categorized into four disability grades with higher scores indicating greater disability: ''Grade I - Little to no disability'' for 0 to 5 days, ''Grade II - Mild disability'' for 6 to 10 days, ''Grade III - Moderate disability'' for 11 to 20 days and ''Grade IV - Severe disability'' for 21 days and over.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Lachaine, Principal Investigator — PeriParm inc.
Locations (1):
- PROxy Network, an initiative of PeriPharm inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No